CLINICAL TRIAL: NCT06704802
Title: Observational Cohort Study Evaluating the Effectiveness of an Education Program (NGAYDAUTIEN) in Combination With Gliclazide MR in the Management of Uncontrolled Type 2 Diabetic Patients.
Acronym: EDUDIA
Status: Completed | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-05762-006
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes
Keywords: observational; HbA1c; type 2 diabetes; Diamicron® MR 60; T2D; patient educational program
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diamicron® MR 60 (originator product) plus educational program: uncontrolled patients with T2D who will be initiated to Diamicron® MR 60 (originator product) plus an educational program
- other OAD except Diamicron®: uncontrolled patients with T2D who will be initiated other OAD except Diamicron®

SUMMARY:
The primary objective is to assess the change of HbA1c level from baseline after a 6-month follow up among uncontrolled patients with T2D who will be initiated to Diamicron® MR 60 (originator product) plus an educational program (NGAYDAUTIEN) as monotherapy or in add on to metformin in comparison to an initiation of an Oral Antidiabetic Drug (OAD) (except Diamicron®) as monotherapy or in add on to metformin.

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 18 years (without upper limit of age)
2. HbA1c value is required at the baseline visit
3. Patients with diagnosis of uncontrolled T2D
4. Initiation of a new OAD as monotherapy or on top of metformin
5. Patient follow-up within the scope of the current medical practice and in the same health center during the 6-month period.

Exclusion Criteria:

1. Diagnosis of diabetes other than T2D
2. HbA1c value not available at baseline
3. Patients who previously attended to the NDT educational program for T2D management
4. Required at baseline an insulin therapy according to national guideline
5. Used any other OAD (except metformin)
6. Used a single pill combination in addition to the medicine of interest
7. Have a severe disease (i.e. cirrhosis, end stage renal disease…)
8. Are unlikely to cooperate in the study or to follow the educational program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female who have a diagnosis of uncontrolled T2D and who initiate a new OAD monotherapy or on top of metformin
Sampling Method: Non-Probability Sample
Enrollment: 678 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
change of HbA1c level (measured in %) from baseline after a 6-month follow-up among the 2 arms | from baseline to 6-month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Servier Affaires Médicales, Suresnes, France

IPD SHARING:
Plan to Share IPD: No